CLINICAL TRIAL: NCT04882514
Title: A Randomized Double Blinded Within Dose, Controlled, Safety and Immunogenicity Study of GAS Vaccine Candidate in Healthy Individuals.
Brief Title: A Trial of a Peptide-based Group A Streptococcal (GAS) Vaccine Candidate in Healthy Individuals.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Griffith University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00089919
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Group A Streptococcal Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Intervention Model Description: Stage 1: The investigators will verify the immediate safety of the J8-K4S2 and p*17-K4S2 vaccines using a test dose in 10 volunteers.
  If there are no safety concerns following the Stage 1 challenge, the study will proceed to a phase 2 double-blind randomized clinical trial. The Rabavert vaccine will be used as a comparator against the 2 investigational arms.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccine p*17-K4S2 (50 µg/mL) Vaccine (Experimental): To evaluate the safety and immunogenicity of p*17-CRM197 (25µg) + K4S2-CRM197 (6.25µg): TOTAL 31.25 µg
  Interventions: Biological: p*17-K4S2
- J8-K4S2 (100 µg/mL ) Vaccine (Experimental): To evaluate the safety and immunogenicity J8-CRM197 (50µg) + K4S2-CRM197 (6.25µg): TOTAL 56.25 µg
  Interventions: Biological: J8-K4S2
- Rabavert Vaccine (Sham Comparator): Comparator vaccine (RABAVERT)
  Interventions: Biological: Rabavert vaccine

INTERVENTIONS:
Biological: p*17-K4S2 — Administer p*17-K4S2 25 μg vaccine at 0, 3, and 6 weeks and evaluate the safety and antibody levels for a total of 6 months after the last injection. All vaccines will be administered intramuscularly
  Arms: Vaccine p*17-K4S2 (50 µg/mL) Vaccine
Biological: J8-K4S2 — Administer a vaccination schedule of J8-K4S2 50μg vaccine at 0, 3, and 6 weeks and evaluate the safety and antibody levels for a total of 6 months after the last injection. All vaccines will be administered intramuscularly
  Arms: J8-K4S2 (100 µg/mL ) Vaccine
Biological: Rabavert vaccine — Administer the standard Rabavert vaccine at 0, 3, and 6 weeks and evaluate the safety and antibody levels for a total of 6 months after the last injection. All vaccines will be administered intramuscularly. The Rabavert vaccine will be used as a control comparator as it has a similar approved dosing schedule to the investigational vaccines.
  Arms: Rabavert Vaccine

SUMMARY:
The purpose of this study is to investigate the safety and antibody (germ fighters) response of experimental (investigational) vaccine candidates against the germ group A streptococcus when injected into the arm of healthy adults.

DETAILED DESCRIPTION:
Group A streptococcus (GAS) is a bacteria that cause a number of different infections that range from mild illnesses to deadly diseases. It is estimated 500,000 deaths occur worldwide each year from GAS. To address these high rates of disease, the investigators want to test a new potential vaccine for safety and immune response in healthy participants.

The investigators will verify the immediate safety of the J8-K4S2 and p*17-K4S2 vaccines using a test dose in 10 volunteers. With respect to J8-K4S2 vaccine, safety of one of the peptide components (J8) has previously been established. Therefore, The investigators will begin with a test dose of J8-K4S2. The first IM injection of J8-K4S2 will be administered to the first participant. The investigators will wait two days, assess safety, then administer J8-K4S2 to a second participant. The investigators will wait two days, assess safety, then administer J8-K4S2 to a third participant. This process will continue until 5 participants have received a test dose of J8- K4S2. If there are no safety concerns with the first 5 participants, the investigators will have shown the preliminary safety of the K4S2 component. If the J8-K4S2 vaccine is well-tolerated, second and third doses of J8-K4S2 will be administered at 3 and 6 weeks, testing the safety of repeated dosing.

The investigators will next administer p*17-K4S2 to a sixth participant, wait two days, assess safety, and administer p*17-K4S2 to a seventh participant. The investigators will wait two days, assess safety, then administer p*17-K4S2 to an eighth participant. This process will continue until 5 participants have received a test dose of p*17-K4S2. If there are no safety concerns, the investigators will have shown the preliminary safety of the p*17 component. If the p*17-K4S2 peptide vaccine is well-tolerated, second and third doses of p*17-K4S2 will be administered at 3 and 6 weeks, testing the safety of repeated dosing.

Following this stage 1 challenge, if no safety concerns arise, the study will proceed to stage 2, with randomized allocation to each arm for 20 more participants who will receive J8-K4S2 vaccine (n=5), p*17-K4S2 vaccine (n=5), and 10 who receive comparator (rabies) vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the purpose and the procedures involved in this study and sign the informed consent form.
* Male or non-pregnant female adults, 18-45 years of age inclusive.
* Non-smoker and in good general health, as determined by medical screening evaluation, performed by PI or delegated sub-investigator no greater than 28 days before the first dose in the form of medical history, clinical laboratory tests and physical examination.
* Normal Electrocardiogram (ECG).
* Echocardiogram (ECHO) that is normal or with findings that are considered trivial and clinically insignificant such as 'Clinically insignificant/trivial mitral regurgitation
* Women must agree not to become pregnant during the trial. If they are sexually active, they must use an effective method of birth control, e.g. insertable, injectable, transdermal, or combination oral contraceptive approved by Health Canada combined with a barrier contraceptive and have negative results on a serum or urine pregnancy test done before administration of study medication.
* Intention to reside in the geographical area for next 10 months and not intending to travel overseas for at least 30 days following the last study vaccine administration.
* Agree not to participate in any other clinical trial during the trial.
* Agree not to donate blood for the duration of the trial.
* Agree to restrain from intensive physical exercise i.e. exercise that varies significantly from an everyday exercise routine, 3 days before and after (± 3 days) administration of each dose, including each interim visit for blood sample collection.
* Up to date on seasonal influenza vaccine and recommended COVID-19 vaccines and booster doses at the time of study enrolment.

Exclusion Criteria:

1. Personal or family history of post-streptococcal disease (rheumatic fever or glomerulonephritis), or collagen-vascular disease
2. Evidence of increased cardiovascular disease risk (defined as >10%, 10- year risk using Framingham score - see Appendix 5). Risk factors include sex, age, systolic blood pressure (mm Hg), smoking status, body mass index (BMI, kg/m2), reported diabetes status and blood pressure
3. Previous use of phentermine (appetite suppressant of the amphetamine and phenethylamine class), fenfluramine or dexfenfluramine known as Fen-Phen, anti-obesity medications (possible association with cardiac valvular abnormalities);
4. Clinical diagnosis or evidence of recent group A streptococcal infection as measured by anti-streptolysin O or anti-DNase B levels exceeding 200 units;
5. Positive group A streptococcus throat culture at screening or rapid antigen test on day of study product administration;
6. Presence of significant acute infection requiring systemic antibiotic treatment within the 14 days prior to each product administration;
7. Pregnant or breast feeding (all women will have a negative pregnancy test result prior to each study product administered);
8. Immunized or intent to immunize with any vaccine or investigational agents within 30 days prior to enrolment through to 30 days following the last study vaccine administration, with the exception of licensed inactivated influenza vaccines and COVID-19 vaccines;
9. Past significant reaction following any previous vaccination;
10. History of hypersensitivity to any diphtheria toxoid or CRM197 containing vaccine;
11. Presence of acute infectious disease or fever (e.g., sub-lingual temperature 38.5°C) within the five days prior to study product administration;
12. Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immunodeficiencies), insulin dependent diabetes, progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, psoriasis, rheumatoid arthritis, asthma, epilepsy or obsessive-compulsive disorder, skin carcinoma excluding non-spreadable skin cancers such as basal cell and squamous cell carcinoma;
13. Evidence and any history of leukaemia, lymphoma, or neoplasm;
14. Presence or suspicion of impaired immune system function. Currently receiving or having within the past three years received immunosuppressive therapy, including systemic steroids, ACTH or inhaled steroids in dosages that are associated with hypothalamic-pituitary-adrenal axis suppression, such as 1mg/kg/day of prednisone or its equivalent or chronic use of inhaled high potency corticosteroids [budesonide 800 µg per day or fluticasone 750 µg];
15. Received blood, blood products or a parenteral immunoglobulin preparation in the past 12 weeks;
16. Evidence of bleeding diathesis or any condition that may be associated with a prolonged bleeding time;
17. Known inherited genetic anomaly (known as cytogenic disorders) e.g., Down's syndrome;
18. Evidence of any condition that, in the opinion of the clinical investigator, might interfere with the evaluation of the study objectives or pose excessive risks to participants;
19. Findings of definite, probable, or possible rheumatic heart disease (RHD), definite or probable acute rheumatic fever (ARF).
20. Inadequate echocardiographic windows for assessment.
21. Echocardiographic findings such as: Cardiac Chambers: left ventricular dilatation (based on LV diameter > 29mm/m2 to BSA); left ventricular dysfunction (Ejection Fraction < 50%; left ventricular hypertrophy (LV wall thickness > 11mm); Right ventricular dysfunction or dilatation (Subjective assessment);
22. Cardiac Valves/Haemodynamic Findings: Clinically significant mitral regurgitation defined: at the discretion of the cardiologist and/or effective regurgitant orifice area of >10mm2; Any degree of valvular stenosis or left ventricular outflow tract obstruction; Pulmonary hypertension (defined as an estimated right ventricular systolic pressure of >30 mmHg, calculated using the peak tricuspid regurgitant jet velocity method);
23. Any aortic regurgitation;
24. Pericardium: greater than trivial pericardial fluid (trivial defined as < 5mm and not circumferential);
25. Pre-existing significant structural valve disease (for example, but not limited to bicuspid aortic valve regardless of haemodynamic effect, mitral valve prolapse regardless of severity of regurgitation, pulmonary stenosis);
26. Other significant congenital lesions (for example, but not limited to aortic coarctation, septal defect, excluding patent foramen ovale (NOTE: findings considered normal developmental variation, specifically including patient foramen ovale and prominent Eustachian valve will not be considered exclusion criteria;
27. Clinical or sub-clinical acute post-streptococcal glomerulonephritis (APSGN),
28. Clinically significant abnormal laboratory results e.g., CBC with differential and platelets, AST, ALT, creatinine, fasting blood sugar, electrolytes (including sodium, potassium, chloride, and bicarbonate);
29. The participant has a diagnosis of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis;
30. The participant has been hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others;
31. The participant is receiving psychiatric drugs but their psychiatric conditions is not stabilized. Participants who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study; *aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate. This is not an absolute contra-indication and clinician judgment will be used to assess the likelihood that this will compromise trial participation and follow-up.
32. The participant has a history of alcohol or drug abuse in the 5 years prior to enrollment. This is not an absolute contra-indication and clinician judgment will be used to assess the likelihood that this will compromise trial participation and follow-up.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 6 months after last dose of vaccine is administered
  Safety is the primary outcome, and will be measured by assessing the clinical symptoms and signs at each study visit and completing standard lab parameters (hematological and biochemical) as well as performing echocardiograms to assess for mitral regurgitation

SECONDARY OUTCOMES:
Immunogenicity | 6 months after last dose of vaccine is administered
  Antibody titre levels will be measured prior to each vaccine dose administered as well as 2 after the last dose and 6 months after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Meier-Stephenson, MD, PhD, Principal Investigator — University of Alberta; Michael Good, MD, PhD, Principal Investigator — Griffith University; Michael Houghton, PhD, Principal Investigator — University of Alberta; Lorne Tyrrell, MD PhD, Principal Investigator — University of Alberta; Michael Hawkes, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Meier-Stephenson V, Hawkes MT, Burton C, Calcutt A, Davis C, Dooley J, Good M, Houghton M, Keeffe E, Kim K, Lepletier A, O'Neil C, Ogbuehi I, Ozberk V, Pandey M, Reynolds S, Seth A, Stokes W, Tse-Chang A, Tyrrell B, Tyrrell DL, Tyrrell GJ, Yaskina M. A phase 1 randomized controlled trial of a peptide-based group A streptococcal vaccine in healthy volunteers. Trials. 2024 Nov 19;25(1):781. doi: 10.1186/s13063-024-08634-4. PMID 39563457